CLINICAL TRIAL: NCT06121401
Title: A Phase IV Trial to Confirm the Efficacy of Olaparib in Combination With Bevacizumab as Frontline Treatment of HRD Positive Ovarian Tumors
Brief Title: First Line Treatment With Olaparib in Combination With Bevacizumab in HRD Positive Patients
Acronym: IOLANTHE
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRFMN-OVA-8542
Record Dates: First submitted 2023-10-23; First posted 2023-11-07 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Carcinoma, Ovarian Epithelial
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — olaparib; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Olaparib - Bevacizumab (Other): Olaparib 300 mg 2*daily + Bevacizumab 15mg/kg (q3w)
  Interventions: Drug: Olaparib; Drug: Bevacizumab

INTERVENTIONS:
Drug: Olaparib — Olaparib is considered the study treatment. Olaparib tablets will be taken at the dose of 300 mg (2 x 150 mg tablet) twice daily adding to bevacizumab at a dose of 15 mg per kilogram of body weight every 3 weeks
  Other Names: Lynparza
Drug: Bevacizumab — Bevacizumab will be taken at a dose of 15 mg per kilogram of body weight every 3 weeks

SUMMARY:
The goal of this prospective, phase IV, multi-centre clinical trial is to to define the proportion of patients with advanced high grade epithelial ovarian cancer (EOC) HRD-positive who will be treated at first line with olaparib in combination with bevacizumab as maintenance and to describe their clinical and demographic characteristics. Other primary objective is to confirm, in a setting close to clinical practice, the efficacy of olaparib concomitant with bevacizumab as maintenance treatment after first-line chemotherapy in patients with advanced high grade EOC HRD-positive and who have received bevacizumab in combination with chemotherapy.

DETAILED DESCRIPTION:
This phase IV study will include two translational research projects:

1. The analyses of the circulating-tumor DNA (ctDNA) derived from plasma samples collected at different time points (liquid biopsy). This sub-study has the aim to evaluate and monitor, through the Next Generation Sequencing approach, the evolution of the disease and the changes in the mutational status of HR-related genes which could lead to different PARPi sensitivity (Translational study no.1).
2. The generation of organotypic models that include cancer stem cells to compare the response of these cancer stem cells to that of bulk tumor cells. This approach will be hopefully able to predict the response to PARPi in ovarian cancer patients. (Translational study no.2)

ELIGIBILITY:
Inclusion Criteria:

1. Patient who has completed first line platinum-taxane chemotherapy
2. Patient on treatment with bevacizumab (patient must have received at least 1 cycle of bevacizumab in combination with chemotherapy). Bevacizumab treatment should have been administered at a dose of 15mg/kg q3 weeks.
3. Patient must be without evidence of disease (NED) or in complete response (CR) or partial response (PR) from her first line treatment.
4. Patients with histologically confirmed high-grade epithelial ovarian, fallopian tube or primary peritoneal cancer and HRD-positive tumor according to the Myriad Mychoice CDx Plus evaluation.
5. Patients must have normal organ and bone marrow function values measured within 28 days before administration of olaparib
6. Normal blood pressure (BP) or adequately treated and controlled hypertension (systolic BP ≤ 140 mmHg and/or diastolic BP ≤ 90 mmHg

8. Patients must have a life expectancy ≥ 16 weeks. 9. Postmenopausal or evidence of non-childbearing status for women of childbearing potential: negative urine or serum pregnancy test within 28 days of olaparib administration and confirmed the day of treatment start.

Exclusion Criteria:

1. Persistent toxicities (Common Terminology Criteria for Adverse Event (CTCAE) grade 2) caused by previous cancer therapy, excluding alopecia
2. Patients with myelodysplastic syndrome/acute myeloid leukaemia or with features suggestive of MDS/AML.
3. Patients with symptomatic uncontrolled brain metastases. A scan to confirm the absence of brain metastases is not required
4. Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection.
5. Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
6. Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV).
7. Patients with known active hepatitis (i.e. Hepatitis B or C).
8. Any previous treatment with PARP inhibitor, including Olaparib.
9. Patients receiving any systemic chemotherapy or radiotherapy (except for palliative reasons) within 3 weeks prior to olaparib.
10. Major surgery within 2 weeks of starting olaparib and patients must have recovered from any effects of any major surgery
11. Administration of other simultaneous chemotherapy drugs, any other anticancer therapy or anti-neoplastic hormonal therapy, or simultaneous radiotherapy during the trial treatment period (hormonal replacement therapy is permitted as are steroidal antiemetics).
12. Concomitant use of known strong CYP3A inhibitors
13. Concomitant use of known strong (eg. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate CYP3A inducers
14. Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT).
15. Patients with a known hypersensitivity to olaparib or any of the excipients of the product.
16. Evidence of any other disease, metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of olaparib or puts the patient at high risk for treatment-related complications.
17. Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements.
18. Breast feeding and pregnant women

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2027-03-15 (Estimated); Study Completion 2027-09-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients treated with olaparib | 42 months
  Define the proportion of patients with advanced high grade epithelial ovarian cancer (EOC) HRD-positive who will be treated at first line with olaparib in combination with bevacizumab as maintenance and to describe their clinical and demographic characteristics
Efficacy of olaparib | 42 months
  Confirm, in a setting close to clinical practice, the efficacy of olaparib concomitant with bevacizumab as maintenance treatment after first-line chemotherapy in patients with advanced high grade EOC HRD-positive and who have received bevacizumab in combination with chemotherapy. The efficacy will be evaluated in terms of PFS rate at 24 months. PFS will be defined as the time from the start of olaparib therapy until disease progression or death whichever comes first

CONTACTS AND LOCATIONS:
Overall Officials: Federica Tomao, Principal Investigator — Università degli Studi di Roma "La Sapienza", Viale del Policlinico 155, Roma
Locations (2):
- Italy (2):
  - Azienda Socio Sanitaria Territoriale (ASST) Lariana, San Fermo della Battaglia, Como
  - Istituto Oncologico Veneto IRCCS, Padua, Italy